CLINICAL TRIAL: NCT02480504
Title: Effects of a 5:2 Diet on Weight Loss and Cardiovascular Risk Factors in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tine Mejlbo Sundfør, MS in Nutrition, ph-D-student, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/1702 (REK); 1702 (Other: REK (The national commitees for research ethics in Norway))
Record Dates: First submitted 2015-06-03; First posted 2015-06-24 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2016-09

CONDITIONS: Obesity; CVD; Dietary Modification
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intermittent energy restriction (Experimental): dietary intervention, intermittent energy restriction. Participants in the experimental group will follow av 5:2 diet and consume a very low calorie diet providing 400 (females) to 600 (males) calories of energy to days a week and for an average male participant, this will reduce energy intake approximately 22%.
  Interventions: Other: dietary intervention intermittent energy restriction
- continuous energy restriction (Active Comparator): dietary intervention, continuous energy restrictions.Participants in the active comparator group will be asked to reduce daily energy intake by 22-23%
  Interventions: Other: continuous energy restriction

INTERVENTIONS:
Other: dietary intervention intermittent energy restriction — Randomized clinical trial
  Arms: intermittent energy restriction
Other: continuous energy restriction
  Arms: continuous energy restriction

SUMMARY:
A randomized clinical trial comparing the effect on weight reduction and cardiometabolic risk factors of intermittent energy restriction and a isocaloric continuous energy restriction in obese subjects.

DETAILED DESCRIPTION:
Background: The optimal diet for treating obesity and cardiovascular disease (CVD) risk is still not clarified. Could a five plus two diet, a form of intermittent energy restriction lead to good adherence, similar weight loss and reduction in CVD risk factors as a isocaloric continuous energy restrictions in obese subjects.

Methods: The study is a randomized controlled clinical trial in 120 men and women between 21 to 70 years with BMI (BMI 30-45 kg/m2), stable weight within ±3 kg last 3 months and 1 additional metabolic syndrome risk component.

Dietary intervention: Randomization will be to one of two diet groups. Participants in the intervention group will follow av 5:2 diet and participants in the control group will follow an isocaloric continuous energy restriction.

Primary research question: Compare the effect on weight reduction of intermittent energy restriction and a isocaloric continuous energy restriction in obese subjects? Secondary research questions Compare the effect of intermittent energy restriction and an isocaloric continuous energy restriction on cardiometabolic risk factors and tolerability and safety in obese subjects. The project consist of to randomized controlled clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 21 to 70 years.
* BMI (BMI 30-45 kg/m2).
* stable weight within ±3 kg last 3 months.
* 1 additional metabolic syndrome risk component.

Exclusion Criteria:

* Diabetes if treated with insulin or incretin analogues.
* History of bariatric surgery.
* Use of antiobesity drugs or supplements.
* Eating disorder.
* Psychiatric illness that contributes to difficulties with study procedures.
* Alcohol or drug abuse.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-09; Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
weight reduction | 1 year
  Compare the effect on weight reduction of intermittent energy restriction and a isocaloric continuous energy restriction in obese subjects

SECONDARY OUTCOMES:
cholesterol | 1 year
  Compare the effect of intermittent energy restriction and isocaloric contiuous energy restriction on cholesterol
adverse events | 1 year
  Compare the effect of intermittent energy restriction and an isocaloric continuous energy restriction on cardiometabolic risk factors and tolerability and safety in obese subjects
blood pressure | 1 year
  Compare the effect of intermittent energy restriction and isocaloric continuous energy restriction on blood pressure
fasting glucose | 1 year
  Compare the effect of intermittent energy restriction and isocaloric continuous energy restriction on fasting glucose
triglycerides | 1 year
  Compare the effect of intermittent energy restriction and isocaloric contiuous energy restriction on fasting triglycerides
HbA1c | 1 year
  Compare the effect of intermittent energy restriction and isocaloric contiuous energy restriction on HbA1c
C-reactive protein (CRP) | 1 year
  Compare the effect of intermittent energy restriction and isocaloric contiuous energy restriction on CRP

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo Universitetssykehus, Ullevål, avdeling for preventiv kardiologi, Oslo, Norway

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Sundfor TM, Svendsen M, Tonstad S. Effect of intermittent versus continuous energy restriction on weight loss, maintenance and cardiometabolic risk: A randomized 1-year trial. Nutr Metab Cardiovasc Dis. 2018 Jul;28(7):698-706. doi: 10.1016/j.numecd.2018.03.009. Epub 2018 Mar 29. PMID 29778565